CLINICAL TRIAL: NCT03554863
Title: Does Optiflow Anesthesia Allow Anethesia Induction "Without Hands" ?
Brief Title: High Flow Oxygen in Patients Undergoing Surgery Under General Anesthesia
Acronym: OPTIFLOW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CMC Ambroise Paré (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017/01
Record Dates: First submitted 2018-05-15; First posted 2018-06-13 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2018-09

CONDITIONS: Anesthesia
Keywords: Anesthesia genral, Oxygen

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Facial mask (Active Comparator)
  Interventions: Device: Facial Mask
- Optiflow anesthesia (Experimental)
  Interventions: Device: Nasal High Flow Oxygen

INTERVENTIONS:
Device: Nasal High Flow Oxygen — Nasal High Flow Oxygen using Optiflow device of Fisher and Paykel
  Arms: Optiflow anesthesia
Device: Facial Mask — Preoxygenation with facial mask
  Arms: Facial mask

SUMMARY:
Preoxygenation remains an important determinant of morbidity and mortality in anesthesia despite advances in mask ventilation and difficult intubation management.

1. The usual practice Preoxygenation prior to the injection of the anesthetic agents is the administration of pure oxygen to delay the occurrence of hypoxemia during the apnea phase and intubation maneuvers. It consists of applying a mask on the patient's face and allowing it to ventilate, ensuring a perfect seal of the device. The end of oxygen exhalation fraction is a good reflection of the alveolar oxygenation and a value of 95% corresponds to a "total" alveolar oxygenation. When this value is reached, the injection of the anesthetic agents (hypnotic, morphine and myorelaxant) leads to the loss of consciousness and apnea, which forces to continue the manual ventilation to the mask. Intubation is performed when the myorelaxation is complete.
2. Anesthetic induction "without the hands" The Optiflow Anesthesia (Fisher and Paykel Healthcare, Auckland, New Zealand) device provides heated, Humidified High-Flow Nasal Oxygen.

The hypothesis of this study is that Humidified High-Flow Nasal Oxygen, should allow anesthetic induction without having to impose the patient the establishment of a facial mask for several minutes before anesthetic induction and the doctor anesthetist assisted ventilation with the mask before intubation.

ELIGIBILITY:
Inclusion Criteria:

* Consent for participation
* Affiliation to the french social security system
* Patients benefit general anesthesia with oral intubation

Exclusion Criteria:

* Pregnant or breastfeeding patients;
* Patients with difficulty of ventilation by Optiflow AnesthesiaTM (facial trauma);
* Patients under the protection of justice
* Patients with drained or undrained pneumothorax;
* Patients with a predicted difficulty of mask ventilation or intubation according to the clinical examination prior to inclusion (arne score ≥ 11) or when treating the patient in the operating room;
* Patients with coronary heart disease, heart failure or respiratory failure;
* Patients with intracranial pathology; patients with arterial oxygen saturation <95% in the open air;
* Patients for whom the surgical procedure requires the installation of a double-lumen tube;
* Patients requiring rapid sequence induction; patients for whom the induction can not be carried out by the sequence sufentanil, propofol, rocuronium;
* Patients with sugammadex allergy;
* Patients placed under judicial protection
* Patients who have already been included in the study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-11-21 (Actual); Primary Completion 2019-02-14 (Actual); Study Completion 2019-02-14 (Actual)

PRIMARY OUTCOMES:
Recourse to another ventilation technique | During the preoxygenation-induction-intubation period (30 min)
  The preoxygenation-induction-intubation period is filmed (audio and video recording) and the use of mask ventilation will be confirmed a posteriori from the audio / video recording by two reviewers.

CONTACTS AND LOCATIONS:
Overall Officials: FISCHLER Marc, MD, Study Chair — Hôpital FOCH
Locations (2):
- France (2):
  - CMC Ambroise Paré, Neuilly-sur-Seine, Île-de-France Region
  - Hôpital Foch, Suresnes, Île-de-France Region

IPD SHARING:
Plan to Share IPD: No